CLINICAL TRIAL: NCT05331261
Title: The Effect of Post-Surgery Exercise in Patients With Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alev Keskin (Other)
Responsible Party: Sponsor-Investigator, Alev Keskin, Co-investigator, Cukurova University
Organization: Cukurova University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ARKeskin
Record Dates: First submitted 2022-04-10; First posted 2022-04-15 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative
Keywords: Ameliyat sonrası ağrıdan nefes egzersizleri.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The Effect of 4-7-8 Breathing Technique on Pain (Experimental): Impact of the 4-7-8 Breathing Technique on Postoperative Pain Following Total Knee Arthroplasty
  Interventions: Procedure: Total diz replacement ameliyatı

INTERVENTIONS:
Procedure: Total diz replacement ameliyatı — Breath exercises

SUMMARY:
postoperative pain; It is acute pain that begins with surgical trauma and decreases during tissue healing. Although it is predictable and treatable, it still seems to be an important problem today. Many researchers in the literature have reported that approximately 50-70% of patients receive inadequate pain treatment after surgery, and many patients complain of moderate or severe pain. Poor control of postoperative pain may cause deep venous thrombosis and delayed wound healing, increased hospital stay, and delayed return to daily life activities. This may negatively affect the quality of life and recovery of patients Therefore, there is a need for methods that increase pain control, such as non-pharmacological methods, to accelerate postoperative recovery. Nurses in postoperative pain management; they help control pain with non-pharmacological methods such as breathing exercises, positioning, relaxation techniques, massage, listening to music, hot application, cold application, and distraction.

DETAILED DESCRIPTION:
This study was designed as a quasi-experimental study to examine the effect of breathing exercise on pain in patients undergoing Total Knee Replacement surgery. This exercise is utterly simple, takes almost no time, requires no equipment and can be done anywhere. Although you can do the exercise in any position, sit with your back straight while learning the exercise. Place the tip of your tongue against the ridge of tissue just behind your upper front teeth, and keep it there through the entire exercise. You will be exhaling through your mouth around your tongue; try pursing your lips slightly if this seems awkward.

* Exhale completely through your mouth, making a whoosh sound.
* Close your mouth and inhale quietly through your nose to a mental count of four.
* Hold your breath for a count of seven.
* Exhale completely through your mouth, making a whoosh sound to a count of eight.
* This is one breath. Now inhale again and repeat the cycle three more times for a total of four breaths.

This study was designed as a quasi-experimental study to examine the effect of breathing exercise on pain in patients undergoing Total Knee Replacement surgery. Note that you always inhale quietly through your nose and exhale audibly through your mouth. The tip of your tongue stays in position the whole time. Exhalation takes twice as long as inhalation. The absolute time you spend on each phase is not important; the ratio of 4:7:8 is important. If you have trouble holding your breath, speed the exercise up but keep to the ratio of 4:7:8 for the three phases. With practice you can slow it all down and get used to inhaling and exhaling more and more deeply.

This exercise is a natural tranquilizer for the nervous system. Unlike tranquilizing drugs, which are often effective when you first take them but then lose their power over time, this exercise is subtle when you first try it but gains in power with repetition and practice. Do it at least twice a day. You cannot do it too frequently. Do not do more than four breaths at one time for the first month of practice. Later, if you wish, you can extend it to eight breaths. If you feel a little lightheaded when you first breathe this way, do not be concerned; it will pass.

ELIGIBILITY:
Inclusion Criteria:

* be over the age of 18,

  * Being able to speak Turkish,
  * Does not have any barriers in communication, understanding and comprehension,
  * Not having visual and hearing impairment,
  * Not taking pain medication 60 minutes before or 30 minutes after the intervention,
  * Volunteering to participate in the research,

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
NRS Scale | Bir dakika
  NRS is a unidimensional scale that uses 11 numbers (from 0 to 10) to measure pain intensity.32 The patient is asked to choose the number that best reflects their pain intensity (0=no pain at all, 10= the worst pain).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Çukurova Üniversitesi, Adana, Sarıçam
  - Çukurova Üniversitesi, Adana, University